CLINICAL TRIAL: NCT05148065
Title: Analysis of Relationship Between Depth of Anesthesia by Inhalation Anesthetic and Primitive Electroencephalogram in Children Under Two Years of Age: a Prospective Observational Study
Brief Title: Frequency Analysis of Raw EEG During Sevoflurane Anesthesia in Children Younger Than 2 Years Old
Status: Completed | Type: Observational
Sponsor: Sang-Hwan Ji (Other)
Responsible Party: Sponsor-Investigator, Sang-Hwan Ji, Clinical assistant professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Other Study IDs: 2109-164-1260
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Anesthesia, General; Sevoflurane; Infant
Keywords: Electroenphalography; Frequency analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: BIS — Bispectral index monitoring
Device: PSi — Patient state index monitoring

SUMMARY:
The purpose of this study is to analyze raw electroencephalogram in infants younger than 2 years old undergoing general anesthesia using sevoflurane.

DETAILED DESCRIPTION:
After obtaining an informed consent from one of the parents, patients undergo routine anesthetic induction using sodium thiopental. Bispectral index and patient state index are both monitored simultaneously. Raw electroencephalogram data are transmitted and recorded via a dedicated equipment. Anesthesia is maintained using sevoflurane with end-tidal level of less than 2 minimum alveolar concentration (MAC) adjusted to age. Fentanyl of up to 1 mcg/kg can be administered in case of increased heart rate and mean blood pressure with a degree of 30% of baseline.

During anesthesia, patients' status of sedation is defined as 'maintenance of surgical state of anesthesia (MOSSA)' when the end-tidal concentration of sevoflurane is maintained between 0.7 and 1.3 MAC and mean blood pressure and heart rate is between 80-120% of baseline.

'Emergence' is defined as a 3-minute period in the middle of continuous decrease in end-tidal concentration of sevoflurane in the range of less than 0.7 MAC and finally reaching 0.2 MAC.

Raw electroencephalogram waves are analyzed by distribution of power along frequency bands and compared according to the state of anesthesia or bispectral index / patient state index value.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged between 4 months and 2 years planned to undergo surgery under general anesthesia
* American Society of Anesthesiologists physical status 1 or 2

Exclusion Criteria:

* History of preterm birth (postconceptual age < 32 wks) or history of mechanical ventilation immediately after birth
* Presence of genetic disease or chromosomal abnormality that can affect brain development
* Presence of disease in central nervous system
* History of head trauma or surgery involving head
* History of hypersensitivity to anesthetic drugs
* Intubated or sedated state before induction of anesthesia
* Difficulty in attaching both the bispectral index and patient state index probes to patient's forehead
* Expected operation time of less than 5 minutes

Ages: 4 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients aged between 4 months and 2 years planned to undergo surgery under general anesthesia, whose American Society of Anesthesiologists physical status are 1 or 2
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Frequency analysis | From start of anesthesia to end of anesthesia, less than 24 hours
  Distribution of raw electroencephalogram waves along frequency bands according to state of anesthesia

SECONDARY OUTCOMES:
Prediction probability | From start of anesthesia to end of anesthesia, less than 24 hours
  Prediction probability of bispectral index and patient state index for maintenance of surgical state of anesthesia
Coherence of BIS and PSi | From start of anesthesia to end of anesthesia, less than 24 hours
  Coherence of BIS and PSi for prediction of state of anesthesia
Emergence delirium and frequency analysis | From start of anesthesia to end of anesthesia, less than 24 hours
  Relationship of distribution of electroencephalogram along frequency band at the 'emergence' state and appearance of emergence delirium at the postanesthesia care unit

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Hwan Ji, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown EN, Lydic R, Schiff ND. General anesthesia, sleep, and coma. N Engl J Med. 2010 Dec 30;363(27):2638-50. doi: 10.1056/NEJMra0808281. No abstract available. PMID 21190458
- [Background] Myles PS, Leslie K, McNeil J, Forbes A, Chan MT. Bispectral index monitoring to prevent awareness during anaesthesia: the B-Aware randomised controlled trial. Lancet. 2004 May 29;363(9423):1757-63. doi: 10.1016/S0140-6736(04)16300-9. PMID 15172773
- [Background] Soehle M, Ellerkmann RK, Grube M, Kuech M, Wirz S, Hoeft A, Bruhn J. Comparison between bispectral index and patient state index as measures of the electroencephalographic effects of sevoflurane. Anesthesiology. 2008 Nov;109(5):799-805. doi: 10.1097/ALN.0b013e3181895fd0. PMID 18946290
- [Background] Soehle M, Kuech M, Grube M, Wirz S, Kreuer S, Hoeft A, Bruhn J, Ellerkmann RK. Patient state index vs bispectral index as measures of the electroencephalographic effects of propofol. Br J Anaesth. 2010 Aug;105(2):172-8. doi: 10.1093/bja/aeq155. Epub 2010 Jun 29. PMID 20587537
- [Background] Koch S, Stegherr AM, Morgeli R, Kramer S, Toubekis E, Lichtner G, von Dincklage F, Spies C. Electroencephalogram dynamics in children during different levels of anaesthetic depth. Clin Neurophysiol. 2017 Oct;128(10):2014-2021. doi: 10.1016/j.clinph.2017.07.417. Epub 2017 Aug 9. PMID 28837907
- [Background] Tokuwaka J, Satsumae T, Mizutani T, Yamada K, Inomata S, Tanaka M. The relationship between age and minimum alveolar concentration of sevoflurane for maintaining bispectral index below 50 in children. Anaesthesia. 2015 Mar;70(3):318-22. doi: 10.1111/anae.12890. Epub 2014 Oct 1. PMID 25271891
- [Background] Cornelissen L, Kim SE, Purdon PL, Brown EN, Berde CB. Age-dependent electroencephalogram (EEG) patterns during sevoflurane general anesthesia in infants. Elife. 2015 Jun 23;4:e06513. doi: 10.7554/eLife.06513. PMID 26102526
- [Background] Kim J, Lee HC, Byun SH, Lim H, Lee M, Choung Y, Kim E. Frontal electroencephalogram activity during emergence from general anaesthesia in children with and without emergence delirium. Br J Anaesth. 2021 Jan;126(1):293-303. doi: 10.1016/j.bja.2020.07.060. Epub 2020 Oct 1. PMID 33010926
- [Background] Eagleman SL, Drover CM, Li X, MacIver MB, Drover DR. Offline comparison of processed electroencephalogram monitors for anaesthetic-induced electroencephalogram changes in older adults. Br J Anaesth. 2021 May;126(5):975-984. doi: 10.1016/j.bja.2020.12.042. Epub 2021 Feb 25. PMID 33640118
- [Background] Seo KH, Kim KM, Lee SK, John H, Lee J. Comparative Analysis of Phase Lag Entropy and Bispectral Index as Anesthetic Depth Indicators in Patients Undergoing Thyroid Surgery with Nerve Integrity Monitoring. J Korean Med Sci. 2019 May 27;34(20):e151. doi: 10.3346/jkms.2019.34.e151. PMID 31124327
- [Background] Avidan MS, Zhang L, Burnside BA, Finkel KJ, Searleman AC, Selvidge JA, Saager L, Turner MS, Rao S, Bottros M, Hantler C, Jacobsohn E, Evers AS. Anesthesia awareness and the bispectral index. N Engl J Med. 2008 Mar 13;358(11):1097-108. doi: 10.1056/NEJMoa0707361. PMID 18337600
- [Background] Katoh T, Kobayashi S, Suzuki A, Kato S, Iwamoto T, Bito H, Sato S. Fentanyl augments block of sympathetic responses to skin incision during sevoflurane anaesthesia in children. Br J Anaesth. 2000 Jan;84(1):63-6. doi: 10.1093/oxfordjournals.bja.a013384. PMID 10740549